CLINICAL TRIAL: NCT01136408
Title: Open Label, Randomised Exploratory Dose Response Study in Pharmacodynamics and Safety of BIBR 1048 (110 mg Twice Daily (b.i.d.) and 150 mg b.i.d.) for 12 Weeks in Patients With Non-valvular Atrial Fibrillation in Comparison to Warfarin
Brief Title: A Dose Response Study of Dabigatran Etexilate(BIBR 1048) in Pharmacodynamics and Safety in Patients With Non-valvular Atrial Fibrillation in Comparison to Warfarin
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Boehringer Ingelheim, Study Chair, Boehringer Ingelheim
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1160.49
Record Dates: First submitted 2010-05-19; First posted 2010-06-03 (Estimated); Results first posted 2010-12-17 (Estimated); Last update posted 2014-03-19 (Estimated); Status verified 2014-02

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Dabigatran; Warfarin

ARMS (3):
- Dabigatran etexilate 220 mg daily (Experimental): Dabigatran etexilate 110 mg capsule, twice a day, oral administration
  Interventions: Drug: Dabigatran etexilate
- Dabigatran etexilate 300 mg daily (Experimental): Dabigatran etexilate 150 mg capsule, twice a day, oral administration
  Interventions: Drug: Dabigatran etexilate
- Warfarin (Active Comparator): Dose-adjusted warfarin based on target INR values
  Interventions: Drug: Warfarin

INTERVENTIONS:
Drug: Dabigatran etexilate — Dabigatran etexilate 110 mg capsule, twice a day, oral administration
  Arms: Dabigatran etexilate 220 mg daily
Drug: Dabigatran etexilate — Dabigatran etexilate 150 mg capsule, twice a day, oral administration
  Arms: Dabigatran etexilate 300 mg daily
Drug: Warfarin — Dose-adjusted warfarin based on target INR values
  Arms: Warfarin

SUMMARY:
The primary objective was to evaluate the safety of dabigatran etexilate(BIBR 1048) administered orally at doses of 110 and 150 mg, twice daily, for 12 weeks in patients with non-valvular atrial fibrillation (paroxysmal, persistent or permanent) in comparison with warfarin.

ELIGIBILITY:
Inclusion criteria Inclusion criteria

1. Patients with non-valvular atrial fibrillation (paroxysmal, persistent or permanent)
2. Patients who had additional risk factor for thromboembolism; one or more of the following conditions/events:

   * Hypertension
   * Diabetes mellitus
   * Left-side heart failure
   * A previous ischemic stroke or transient ischemic attack
   * Age 75 years or older
   * A history of coronary artery diseases

Exclusion criteria Exclusion criteria

1. Patients diagnosed as having a valvular heart disease by echocardiography, or patients who had a history of prosthetic valve replacement or valve surgery
2. Patients who were to receive electric defibrillation or pharmacological defibrillation during the study period
3. Patients who developed stroke or transient ischemic attack within 30 days before the date of informed consent
4. Patients who developed myocardial infarction or were admitted to hospital due to acute coronary syndrome or for percutaneous transluminal coronary angioplasty within 3 months before the date of informed consent or patients underwent coronary stenting within 6 months before the date of informed consent
5. Patients with atrial myxoma or left ventricular thrombosis
6. Patients with contraindication to anticoagulant therapies
7. Patients scheduled for major surgery or invasive procedure
8. Patients having major bleeding from non-gastrointestinal organs within 6 months before the date of informed consent
9. Patients with uncontrolled hypertension

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 2005-11; Primary Completion 2006-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (28):
- Japan (28):
  - 1160.49.024 Boehringer Ingelheim Investigational Site, Aki-gun, Hiroshima
  - 1160.49.025 Boehringer Ingelheim Investigational Site, Fukuoka, Fukuoka
  - 1160.49.026 Boehringer Ingelheim Investigational Site, Fukuoka, Fukuoka
  - 1160.49.021 Boehringer Ingelheim Investigational Site, Himeji, Hyogo
  - 1160.49.027 Boehringer Ingelheim Investigational Site, Iizuka,Fukuoka
  - 1160.49.013 Boehringer Ingelheim Investigational Site, Kyoto, Kyoto
  - 1160.49.011 Boehringer Ingelheim Investigational Site, Nagoya, Aichi
  - 1160.49.012 Boehringer Ingelheim Investigational Site, Nagoya, Aichi
  - 1160.49.004 Boehringer Ingelheim Investigational Site, Naka-gun, Ibaragi
  - 1160.49.022 Boehringer Ingelheim Investigational Site, Okayama, Okayama
  - 1160.49.023 Boehringer Ingelheim Investigational Site, Okayama, Okayama
  - 1160.49.006 Boehringer Ingelheim Investigational Site, Oota, Tokyo
  - 1160.49.016 Boehringer Ingelheim Investigational Site, Osaka, Osaka
  - 1160.49.017 Boehringer Ingelheim Investigational Site, Osaka, Osaka
  - 1160.49.018 Boehringer Ingelheim Investigational Site, Osaka, Osaka
  - 1160.49.019 Boehringer Ingelheim Investigational Site, Osaka, Osaka
  - 1160.49.020 Boehringer Ingelheim Investigational Site, Sakai, Osaka
  - 1160.49.001 Boehringer Ingelheim Investigational Site, Sapporo, Hokkaido
  - 1160.49.028 Boehringer Ingelheim Investigational Site, Sapporo, Hokkaido
  - 1160.49.002 Boehringer Ingelheim Investigational Site, Sendai, Miyagi
  - 1160.49.005 Boehringer Ingelheim Investigational Site, Shinjuku, Tokyo
  - 1160.49.014 Boehringer Ingelheim Investigational Site, Suita, Osaka
  - 1160.49.015 Boehringer Ingelheim Investigational Site, Suita, Osaka
  - 1160.49.007 Boehringer Ingelheim Investigational Site, Tokorozawa, Saitama
  - 1160.49.009 Boehringer Ingelheim Investigational Site, Toyama, Toyama
  - 1160.49.003 Boehringer Ingelheim Investigational Site, Tsuchiura, Ibaragi
  - 1160.49.029 Nagano National Hospital, Ueda, Nagano
  - 1160.49.008 Boehringer Ingelheim Investigational Site, Yokohama, Kanagawa

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eight patients were randomised but not treated with study drug, hence resulting in 174 patients as enrolled and 166 who were actually treated.
Period: Overall Study
Arm/Group | Dabigatran Etexilate 220 mg Daily | Dabigatran Etexilate 300 mg Daily | Warfarin
Started | 46 | 58 | 62
Completed | 41 | 49 | 57
Not Completed | 5 | 9 | 5
Not completed — Adverse Event | 4 | 8 | 4
Not completed — Protocol Violation | 1 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dabigatran Etexilate 220 mg Daily | Dabigatran Etexilate 300 mg Daily | Warfarin | Total
Number analyzed (Participants) | 46 | 58 | 62 | 166
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.9 (7.5) | 68.3 (9.1) | 67.4 (8.8) | 68.4 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 5 | 5 | 20
  Male | 36 | 53 | 57 | 146

OUTCOME MEASURES:

1. Primary Outcome: Frequency (Occurrence Rates) of Major Bleeding Event
Description: The percentage of patients with major bleeding event.
  Major bleeding was defined as any bleed fulfilling one of the following conditions:
  * Fatal or life-threatening
  * Retroperitoneal, intracranial, intraocular, or intraspinal bleeding (verified by objective testing)
  * Bleeding requiring surgical treatment
  * Clinically overt bleeding leading to a transfusion (erythrocyte component transfusion or whole blood transfusion) of 4.5 units (equal to 2 units in EU/US) or more
  * Clinically overt bleeding leading to a fall in haemoglobin of at least 2 g/dL
Time Frame: upto 15 weeks
Population: Safety set was used for safety endpoints. Full analysis set was used for efficacy endpoints. The safety set comprises all patients who were treated with trial medication at least once. The full analysis set comprises all patients who were randomised and treated with trial medication at least once. No data was imputed.
Measure: Number; unit: Percentage of patients
Arm/Group | Dabigatran Etexilate 220 mg Daily | Dabigatran Etexilate 300 mg Daily | Warfarin
Number analyzed (Participants) | 46 | 58 | 62
Percentage of patients | 0 | 1.7 | 3.2

2. Primary Outcome: Frequency (Occurrence Rates) of Clinically Relevant Bleeding Event
Description: The percentage of patients with clinically relevant bleeding event.
  Any bleed that did not qualify as a major bleed was defined as a minor bleed; minor bleed which fulfilled one of the criteria below was defined as a clinically relevant bleeding event:
  * A skin haematoma of at least 25 sqcm
  * Spontaneous nose bleed lasting for more than 5 minutes
  * Macroscopic haematuria (either spontaneous or, if associated with an intervention, lasting more than 24 hours)
  * Spontaneous rectal bleeding (more than spotting on toilet paper)
  * Gingival bleeding lasting for more than 5 minutes
  * Bleeding leading to hospitalisation
  * Bleeding leading to blood transfusion (erythrocyte component transfusion or whole blood transfusion) of less than 4.5 units (equal to 2 units in EU/US)
  * Any other bleeding considered clinically relevant by the investigator
Time Frame: upto 15 weeks
Population: as for outcome 1
Measure: Number; unit: Percentage of patients
Arm/Group | Dabigatran Etexilate 220 mg Daily | Dabigatran Etexilate 300 mg Daily | Warfarin
Number analyzed (Participants) | 46 | 58 | 62
Percentage of patients | 4.3 | 8.6 | 8.1

3. Primary Outcome: Frequency (Occurrence Rates) of Nuisance Bleeding Event
Description: The percentage of patients with nuisance bleeding event
  Any bleed that did not qualify as a major bleed was defined as a minor bleed; all minor bleeding events not fulfilling one of the criteria below was defined as a nuisance bleeding event:
  * A skin haematoma of at least 25 sqcm
  * Spontaneous nose bleed lasting for more than 5 minutes
  * Macroscopic haematuria (either spontaneous or, if associated with an intervention, lasting more than 24 hours)
  * Spontaneous rectal bleeding (more than spotting on toilet paper)
  * Gingival bleeding lasting for more than 5 minutes
  * Bleeding leading to hospitalisation
  * Bleeding leading to blood transfusion (erythrocyte component transfusion or whole blood transfusion) of less than 4.5 units (equal to 2 units in EU/US)
  * Any other bleeding considered clinically relevant by the investigator
Time Frame: Upto 15 weeks
Population: as for outcome 1
Measure: Number; unit: Percentage of patients
Arm/Group | Dabigatran Etexilate 220 mg Daily | Dabigatran Etexilate 300 mg Daily | Warfarin
Number analyzed (Participants) | 46 | 58 | 62
Percentage of patients | 19.6 | 29.3 | 19.4

4. Secondary Outcome: Frequency (Occurrence Rates) of a Composite Clinical Endpoint.
Description: Percentage of patients with the composite clinical endpoint (ischemic or haemorrhagic stroke (fatal or non-fatal), transient ischemic attacks, systemic embolism, myocardial infarction (fatal or non-fatal), other major adverse cardiac events, and death)
Time Frame: Upto 15 weeks
Population: as for outcome 1
Measure: Number; unit: Percentage of patients
Arm/Group | Dabigatran Etexilate 220 mg Daily | Dabigatran Etexilate 300 mg Daily | Warfarin
Number analyzed (Participants) | 46 | 58 | 62
Percentage of patients | 0 | 0 | 1.6

5. Secondary Outcome: Frequency (Occurrence Rates) of Ischemic or Haemorrhagic Stroke (Fatal or Non-fatal)
Description: The percentage of patients with ischemic or haemorrhagic stroke (fatal or non-fatal)
Time Frame: Upto 15 weeks
Population: as for outcome 1
Measure: Number; unit: Percentage of patients
Arm/Group | Dabigatran Etexilate 220 mg Daily | Dabigatran Etexilate 300 mg Daily | Warfarin
Number analyzed (Participants) | 46 | 58 | 62
Percentage of patients | 0 | 0 | 1.6

6. Secondary Outcome: Frequency (Occurrence Rates) of Transient Ischemic Attack
Description: The percentage of patients with transient ischemic attack
Time Frame: Upto 15 weeks
Population: as for outcome 1
Measure: Number; unit: Percentage of patients
Arm/Group | Dabigatran Etexilate 220 mg Daily | Dabigatran Etexilate 300 mg Daily | Warfarin
Number analyzed (Participants) | 46 | 58 | 62
Percentage of patients | 0 | 0 | 0

7. Secondary Outcome: Frequency (Occurrence Rates) of Systemic Embolism
Description: The percentage of patients with systemic embolism
Time Frame: Upto 15 weeks
Population: as for outcome 1
Measure: Number; unit: Percentage of patients
Arm/Group | Dabigatran Etexilate 220 mg Daily | Dabigatran Etexilate 300 mg Daily | Warfarin
Number analyzed (Participants) | 46 | 58 | 62
Percentage of patients | 0 | 0 | 0

8. Secondary Outcome: Frequency (Occurrence Rates) of Myocardial Infarction (Fatal or Non-fatal)
Description: The percentage of patients with myocardial infarction (fatal or non-fatal)
Time Frame: Upto 15 weeks
Population: as for outcome 1
Measure: Number; unit: Percentage of patients
Arm/Group | Dabigatran Etexilate 220 mg Daily | Dabigatran Etexilate 300 mg Daily | Warfarin
Number analyzed (Participants) | 46 | 58 | 62
Percentage of patients | 0 | 0 | 0

9. Secondary Outcome: Frequency (Occurrence Rates) of Other Major Adverse Cardiac Events
Description: The percentage of patients with other major adverse cardiac events
Time Frame: Upto 15 weeks
Population: as for outcome 1
Measure: Number; unit: Percentage of patients
Arm/Group | Dabigatran Etexilate 220 mg Daily | Dabigatran Etexilate 300 mg Daily | Warfarin
Number analyzed (Participants) | 46 | 58 | 62
Percentage of patients | 0 | 0 | 0

10. Secondary Outcome: Frequency (Occurrence Rates) of Death
Description: The percentage of patients with death
Time Frame: Upto 15 weeks
Population: as for outcome 1
Measure: Number; unit: Percentage of patients
Arm/Group | Dabigatran Etexilate 220 mg Daily | Dabigatran Etexilate 300 mg Daily | Warfarin
Number analyzed (Participants) | 46 | 58 | 62
Percentage of patients | 0 | 0 | 0

11. Primary Outcome: Incidence and Severity of Adverse Events
Description: Intensity of event is categorised as mild, moderate and severe.
Time Frame: Upto 15 weeks
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Dabigatran Etexilate 220 mg Daily | Dabigatran Etexilate 300 mg Daily | Warfarin
Number analyzed (Participants) | 46 | 58 | 62
participants
  Mild | 28 | 46 | 35
  Moderate | 1 | 1 | 4
  Severe | 0 | 2 | 2

12. Primary Outcome: Discontinuation of the Study Drug Due to Adverse Events
Description: Discontinuation of the study drug due to adverse events.
Time Frame: Upto 15 weeks
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Dabigatran Etexilate 220 mg Daily | Dabigatran Etexilate 300 mg Daily | Warfarin
Number analyzed (Participants) | 46 | 58 | 62
participants | 4 | 8 | 4

13. Secondary Outcome: Anticoagulation Effects Trough aPTT (Activated Partial Thromboplastin Time)
Description: The blood coagulation parameter aPTT was assessed in patients allocated to the dabigatran etexilate groups at week 0, prior to drug administration and at the trough at week 1, 4 and 12.
Time Frame: Week 0,1,4 and 12
Population: Full Analysis Set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: seconds
Arm/Group | Dabigatran Etexilate 220 mg Daily | Dabigatran Etexilate 300 mg Daily
Number analyzed (Participants) | 46 | 58
seconds
  week 0, N=46 , N=58 | 32.4 (12.7) | 34.0 (25.0)
  week 1, N=41, N=55 | 40.2 (16.4) | 45.0 (20.7)
  week 4, N=40, N=50 | 40.9 (16.2) | 45.0 (17.9)
  week 12, N=40, N=48 | 41.8 (17.3) | 44.1 (18.2)

14. Secondary Outcome: Anticoagulation Effects Trough ECT (Ecarin Clotting Time)
Description: The blood coagulation parameter ECT was assessed in patients allocated to the dabigatran etexilate groups at week 0, prior to drug administration and at the trough at week 1, 4 and 12.
Time Frame: Week 0,1,4 and 12
Population: Full Analysis Set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: seconds
Arm/Group | Dabigatran Etexilate 220 mg Daily | Dabigatran Etexilate 300 mg Daily
Number analyzed (Participants) | 46 | 58
seconds
  week 0, N=46 , N=58 | 35.6 (9.39) | 36.3 (10.5)
  week 1, N=41, N=55 | 53.4 (23.5) | 63.2 (35.3)
  week 4, N=40, N=50 | 51.4 (23.1) | 58.9 (27.7)
  week 12, N=40, N=48 | 52.7 (24.1) | 56.9 (28.5)

15. Secondary Outcome: Anticoagulation Effects Trough INR (International Normalised Ratio)
Description: The blood coagulation parameter INR was assessed in patients allocated to the dabigatran etexilate groups at week 0, prior to drug administration and at the trough at week 1, 4 and 12.
Time Frame: Week 0,1,4 and 12
Population: Full Analysis Set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Dabigatran Etexilate 220 mg Daily | Dabigatran Etexilate 300 mg Daily
Number analyzed (Participants) | 46 | 58
ratio
  week 0, N=46 , N=58 | 1.87 (35.7) | 2.03 (33.4)
  week 1, N=41, N=55 | 1.35 (14.0) | 1.49 (20.0)
  week 4, N=40, N=50 | 1.35 (16.6) | 1.46 (18.0)
  week 12, N=39, N=49 | 1.43 (21.2) | 1.49 (25.2)

16. Secondary Outcome: Anticoagulation Effects Trough 11-dehydrothromboxane B2
Description: Analysis based on concomitant use of aspirin compared to no aspirin users. 11-dehydrothromboxane B2 is measured in urine of patients.
Time Frame: Week 0 and 12
Population: Per Protocol Analysis Set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg/mg creatinine
Arm/Group | Dabigatran Etexilate 220 mg Daily | Dabigatran Etexilate 300 mg Daily | Warfarin
Number analyzed (Participants) | 43 | 56 | 58
pg/mg creatinine
  week 0 without aspirin, N=34, N=43, N=37 | 2730 (80.5) | 3190 (65.5) | 3080 (52.3)
  week 0 with aspirin, N=9, N=12, N=20 | 1890 (49.5) | 1480 (49.9) | 1660 (54.3)
  week 12 without aspirin, N=34, N=42, N=37 | 3350 (62.8) | 3430 (56.5) | 3520 (53.9)
  week 12 with aspirin, N=9, N=13, N=21 | 2380 (71.2) | 1830 (30.4) | 1420 (55.3)

17. Secondary Outcome: Steady-state Pharmacokinetics of Total Dabigatran Trough Plasma Concentration
Time Frame: Week 1,4 and 12
Population: Full Analysis Set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Dabigatran Etexilate 220 mg Daily | Dabigatran Etexilate 300 mg Daily
Number analyzed (Participants) | 46 | 58
ng/mL
  week 1, N=41, N=55 | 53.1 (69.0) | 78.1 (75.8)
  week 4, N=40, N=50 | 55.6 (62.5) | 78.2 (68.1)
  week 12, N=39, N=49 | 63.0 (62.1) | 75.1 (63.3)

18. Primary Outcome: Changes in Laboratory Test Values
Description: The number of patients with ALT, AST, alkaline phosphatase, or bilirubin exceeded the upper limit of normal (ULN) range
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Dabigatran Etexilate 220 mg Daily | Dabigatran Etexilate 300 mg Daily | Warfarin
Number analyzed (Participants) | 46 | 58 | 60
participants
  ALT > 1 x ULN | 1 | 4 | 4
  AST > 1 x ULN | 0 | 4 | 5
  Alkaline phosphatase > 1 x ULN | 2 | 3 | 1
  Total bilirubin > 1 x ULN | 6 | 7 | 8

ADVERSE EVENTS:
Time Frame: First administration to end of study
Arm/Group | Dabigatran Etexilate 220 mg Daily | Dabigatran Etexilate 300 mg Daily | Warfarin
Serious Adverse Events (participants affected / at risk) | 0/46 | 6/58 | 5/62
Other Adverse Events (participants affected / at risk) | 9/46 | 25/58 | 16/62
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dabigatran Etexilate 220 mg Daily (N=46) | Dabigatran Etexilate 300 mg Daily (N=58) | Warfarin (N=62)
Pneumonia (Infections and infestations) | 0 | 1 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1
Haemorrhagic cerebral infarction (Nervous system disorders) | 0 | 0 | 1
Atrioventricular block third degree (Cardiac disorders) | 0 | 1 | 0
Cardiac arrest (Cardiac disorders) | 0 | 1 | 0
Cardiac failure (Cardiac disorders) | 0 | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 0 | 1
Muscle fatigue (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Prostatic haemorrhage (Reproductive system and breast disorders) | 0 | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Laryngeal injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dabigatran Etexilate 220 mg Daily (N=46) | Dabigatran Etexilate 300 mg Daily (N=58) | Warfarin (N=62)
Nasopharyngitis (Infections and infestations) | 5 | 10 | 8
Insomnia (Psychiatric disorders) | 1 | 3 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 5 | 3
Diarrhoea (Gastrointestinal disorders) | 1 | 4 | 2
Abdominal pain upper (Gastrointestinal disorders) | 0 | 3 | 0
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 1 | 7 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract